CLINICAL TRIAL: NCT06420401
Title: Precision Treatment of Hyperuricemia Based on Different Combinations of Prebiotics
Brief Title: Prebiotics and the Management of Hyperuricemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Min Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Prebiotics-2024
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Subjects With Hyperuricemia
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dietary supplement: araboxylan (Experimental): Eligilable subjects are instructed to take one pocket of araboxylan during the first week, followed by two pockets of araboxylan during the remaining 11 weeks.
  Interventions: Dietary Supplement: araboxylan
- Dietary supplement: inulin (Experimental): Eligilable subjects are instructed to take one pocket of inulin during the first week, followed by two pockets of inulin during the remaining 11 weeks.
  Interventions: Dietary Supplement: inulin
- Dietary supplement: inulin and araboxylan (Experimental): Eligilable subjects are instructed to take one pocket of inulin and arabosylan during the first week, followed by two pockets of inulin and araboxylan during the remaining 11 weeks.
  Interventions: Dietary Supplement: inulin and araboxylan
- Dietary supplement: placebo (Placebo Comparator): Eligilable subjects are instructed to take one pocket of maltodextrin during the first week, followed by two pockets of maltodextrin during the remaining 11 weeks.
  Interventions: Dietary Supplement: placebo control

INTERVENTIONS:
Dietary Supplement: araboxylan — During the study period, subjects are instructed to take one pocket of arabosylan per day during the first week, followed by two pockets of araboxylan per day during the remianing 11 weeks. Aside from the dietary supplement provided, all participants are instructed to continue their normal routine and not make any changes to their dietary habits or physical activity.
  Arms: Dietary supplement: araboxylan
Dietary Supplement: inulin — During the study period, subjects are instructed to take one pocket of inulin per day during the first week, followed by two pockets of inulin per day during the remianing 11 weeks. Aside from the dietary supplement provided, all participants are instructed to continue their normal routine and not make any changes to their dietary habits or physical activity.
  Arms: Dietary supplement: inulin
Dietary Supplement: inulin and araboxylan — During the study period, subjects are instructed to take one pocket of inulin and araboxylan per day during the first week, followed by two pockets of inulin and araboxylan per day during the remianing 11 weeks. Aside from the dietary supplement provided, all participants are instructed to continue their normal routine and not make any changes to their dietary habits or physical activity.
  Arms: Dietary supplement: inulin and araboxylan
Dietary Supplement: placebo control — During the study period, subjects are instructed to take one pocket of placebo control per day during the first week, followed by two pockets of placebo control per day during the remianing 11 weeks. Aside from the dietary supplement provided, all participants are instructed to continue their normal routine and not make any changes to their dietary habits or physical activity.
  Arms: Dietary supplement: placebo

SUMMARY:
Hyperuricemia is a major risk factor for many chronic diesease. Recently, gut mcirobiota has been identified as a novel theraputic target for hyperuricemia. Both annimal studies and pilot human trials have demonstrated that administration of prebiotics help delay the progression of hyperuricemia throuh several mechanisms. This trial aims to examine its protective effects and potential mechanisms in clinical trials.

DETAILED DESCRIPTION:
Hyperuricemia is a major risk factor for many chronic diseases. Recently, dysbiosis of gut microbiota has been reported to play an important role in the pathogenesis of hyperuricemia. Animal studies have demonstrated that administration of prebiotics help delay the progression of hyperuricemia through several mechanisms such as reduction in endotoxemia, and enhanced production of short-chain fatty acids and hippuric acid.

However, whether administration of prebiotics also has a protective effect in subjects with hyperuricemia remain under-explored. Moreover, whether the original gut microbiota will influence the protective effect of prebiotics remains largely unknown.

ELIGIBILITY:
Inclusion Criteria:

* Local residents aged between 18-80 years old;

  * Stable weight (<5% weight change over the past 3 months);
  * Fsating uric acid > 420 umol/L for male and > 360 umol/L for female on two different days;
  * Not taking uric acid lowering drugs or have stopped taking uric acid lowering drugs for over 4 weeks at the time of recruitment;
  * Absence of any diet or medication that might interfere with uric acid metabolims or gut microbiota, especially antibiotics, prebiotics or probiotics at the least 4 weeks before recruitment

Exclusion Criteria:

* Acute illness or evidence of any acute or chronic inflammatroy of infective diseases;

  * Participation in regular diet program more than 2 times per week in the lastest 3 months prior to recruitment;
  * Mental illness rendering them unable to understand the nature, scope, and possible consequences of the study;
  * Women of childbearing age who are pregant, breast-feeding or preparing for pregnancy; patients who had surgey within the past 6 months or planned surgery during the trial period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of serum uric acid | from baseline to 12 weeks after intervention
  change of fasting uric acid level assessed by biochemical detector
Change of excretion of uric acid | from baseline to 12 weeks after intervention
  excretion rate of uric acid assessed by secretion rate of uric acid in urine during 3 hours

SECONDARY OUTCOMES:
Change of gut microbiota | from baseline to 12 weeks after intervention
  Alterations of the composition of gut microbiota evaluated by metagenomics
Change of microbial metabolites | from baseline to 12 weeks after intervention
  Untargeted metabolomics will be used to assess the alterations of microbial metabolites with high performance liquid chromatography-mass spectrometry
Change in insulin sensitivity | from baseline to 12 weeks after intervention
  HOMA-IR will be used to assess the change of insulin sensitivity
Change in waist circumference | from baseline to 12 weeks after intervention
  change in waist circumference assessed by tape
Change in blood pressure | from baseline to 12 weeks after intervention
  change in blood pressure assessed by electronic sphymomanometer
Change in lipid profiles | from baseline to 12 weeks after intervention
  change in total cholesterol, triglycerides, LDL-c and HDL-c assessed by biochemical detector

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Nutrition and Food Hygiene, Guangzhou, Guangdong
  - Sun Yat-Sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No